CLINICAL TRIAL: NCT05355571
Title: The Impact of Probiotic Supplementation on Antibiotic Induced Changes in Gastrointestinal Function And/or Faecal Microbiota Composition (FANTIB)
Brief Title: The Impact of Probiotic Supplementation on Antibiotic Induced Changes in Gastrointestinal Function And/or Faecal Microbiota Composition
Acronym: FANTIB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cultech Ltd (Industry)
Collaborators: Comac Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: FANTIB
Record Dates: First submitted 2022-04-19; First posted 2022-05-02 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Antibiotic Side Effect

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active (Active Comparator): Participants will consume a probiotic containing lactic acid bacteria and Saccharomyces boulardii at a dose of 35 billion per day for 10 days alongside an oral antibiotic at standard dosage administered for fixed period
  Interventions: Dietary Supplement: LAB4 + Saccharomyces boulardii
- Placebo (Placebo Comparator): Participants will consume a placebo alongside an oral antibiotic at standard dosage administered for fixed period
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: LAB4 + Saccharomyces boulardii — Probiotic containing lactic acid bacteria and Saccharomyces boulardii at a dose of 35 billion per day
  Arms: Active
Dietary Supplement: Placebo — Placebo
  Arms: Placebo

SUMMARY:
To investigate whether probiotic supplementation during the consumption of oral antibiotics can impact gastrointestinal responses and/or the regrowth of the gut microbiota.

DETAILED DESCRIPTION:
The human gut (gastrointestinal tract) is home to more than a trillion mostly "friendly bacteria" = the gut microbiota - that support the well-being and health of an individual through a variety of mechanisms. Antibiotic treatment impacts on the microbiota and reduces the overall numbers and diversity which causes metabolic shifts and increases susceptibility to colonization by potentially pathogenic and/or resistant bacteria and thereby increases the risk of bacterial antibiotic resistance. This trial aims to investigate whether probiotic supplementation during the consumption of oral antibiotics can impact the gastrointestinal responses and/or the composition/functionality of the regrowth of the gut microbiota.

The trial will be a double blinded, placebo-controlled study consisting of 50 participants (25 per group), aged 18-65, to be enrolled after being prescribed a 5 to 10-day course of antibiotics. The study will be randomized through an independent statistician.

The study will involve three site visits, the first visit occurs at enrolment when the participant is randomised and measures of height, body weight and blood pressure are taken. The participants will also answer a quality of life questionnaire at visit 1 and will receive the study intervention. A stool sample will be collected at this visit (if possible) and the participant will be given two more stool sample collection kits, a gastrointestinal tract symptom record sheet too b completed daily throughout the study and a bowel habit diary to be completed per defecation..

The second visit will take place the day after the completion of the prescribed antibiotic course and at this visit participants will return a stool sample collected at home the previous day, and asked to complete another quality of life questionnaire. The final visit will take place at around day 30, when again they will return a stool sample collected within 48 hours of the visit, return all gastrointestinal symptom record sheets and bowel habit diaries as well as returning any unused intervention (for compliance monitoring). Scientists will use the information and samples collected to determine if there was any benefit to taking the probiotic supplement.

It is considered that the daily intake of the probiotics will improve general wellbeing and mental health. Due to the chance that the participant may receive the placebo, it is perceived that these benefits will be confined to the participants who are randomly assigned the intervention. Participation in the study will bring more information and will improve our understanding of the benefits of daily probiotic supplementation.

There have been no adverse reactions associated with the regular consumption of this probiotic product but participants may experience mild side effects such as a change in bowel habit and/ or increased flatulence (intestinal gas) during the first few days of taking the supplement.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged 18-65
2. Receiving a 5 to 10 day course of oral antibiotics
3. Willing to provide 3 faecal samples over the duration of the study
4. Willing to refrain from taking non-GP (general practitioner) prescribed antibiotics

Exclusion Criteria:

1. Consumed regular probiotic supplementation within the last 1 month prior to the study
2. Consumed any antibiotic within the last 3 months
3. Prescribed antibiotics for a gastrointestinal related issue
4. Diagnosed with diabetes
5. Are immunodeficient or undergoing immunosuppressive therapy
6. Diagnosed with arrhythmia, ventricular extrasystole, atrioventricular block or other cardiovascular disease deemed as a risk by study doctor
7. Diagnosed with a cardiovascular disease
8. Pregnancy or planning pregnancy
9. Diagnosed with a severe systemic disease e.g. cancer, dementia, advanced organ failure.
10. Unexplained loss of weight in recent months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-11-18 (Actual); Primary Completion 2023-01-17 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Microbiological analysis of stool samples as a measure of abundance within the microbiota post antibiotic consumption. | One month post antibiotic treatment/ probiotic supplementation
  Stool samples will be streaked out onto specific agar to measure the viable abundance of specific bacteria and fungi including; Lactobacillus, Enterobacteria, Enterococci, Staphylococci, Yeast, Bifidobacteria and Bacteroides. Microbiological counts (Log10 CFU/g(Colony forming unit/g)) will then be analysed and compared.
Next generation sequencing (NGS) analysis of stool samples as a measure of microbiome diversity and abundance within the microbiota post antibiotic consumption. | One month post antibiotic treatment/ probiotic supplementation
  Genomic DNA will be extracted from stool samples and subsequently run through Illumina MiSeq to produce sequencing data which can be used to analyse diversity (Alpha and Beta) changes in the microbiome along with changes in abundance of taxa.

SECONDARY OUTCOMES:
Quality of life questionnaires to measure quality of life post probiotic supplementation | One month post antibiotic treatment/ probiotic supplementation
  Quality of life questionnaires will be completed at the start, post antibiotic treatment and end of study. Questionnaires are rated on a scale from 1 (very poor) to 10 (very good) and questions include; General wellness, state of health, state of energy, state of mood and sleep quality.
Questionnaire of gastrointestinal health to measure gastrointestinal health post probiotic supplementation. | One month post antibiotic treatment/ probiotic supplementation
  A daily gastrointestinal tract symptom record sheet which involves ticking off symptoms is present. Symptoms include; Abdominal pains, Bloating, stomach rumbling, vomiting/nausea, acid regurgitation/heartburn, increased flatulence and increased belching.
Bowel habit diary to measure gastrointestinal health post probiotic supplementation. | One month post antibiotic treatment/ probiotic supplementation
  A bowel habit diary questionnaire to be completed for every attempted bowel motion during the study. Questions include; 1. Were you able to pass a stool?, 2. Did you feel an urgent need to pass the bowel motion?, 3. Did you strain to start the bowel motion?, 4. Were you left with a feeling of incomplete evacuation?, 5. Please rate the appearance of your bowel motion using the bristol stool score (1-7).

CONTACTS AND LOCATIONS:
Overall Officials: Aleksandrina Panteleeva, Principal Investigator — Comac Medical
Locations (1):
- Comac Medical, Sofia, Bulgaria

IPD SHARING:
Plan to Share IPD: No